CLINICAL TRIAL: NCT03950622
Title: A Phase 3, Multicenter, Randomized, Double-blind, Active Comparator-controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of V114 in Healthy Adults 50 Years of Age or Older (PNEU-AGE)
Brief Title: Safety and Immunogenicity of V114 in Healthy Adults (V114-019/PNEU-AGE)
Acronym: PNEU-AGE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V114-019; 2018-004316-22 (Other: EudraCT Number); V114-019 (Other: Merck); 194845 (Registry Identifier: Japic-CTI)
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Results first posted 2021-03-18 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-03

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V114 (Experimental): Single intramuscular (IM) dose at 0.5 mL of V114 pneumococcal conjugate vaccine at Visit 1 (Day 1)
  Interventions: Biological: V114
- Prevnar 13™ (Active Comparator): Single IM dose at 0.5 mL of Prevnar 13™ at Visit 1 (Day 1)
  Interventions: Biological: Prevnar 13®

INTERVENTIONS:
Biological: V114 — 15-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F in each 0.5 mL dose.
  Arms: V114
Biological: Prevnar 13® — 13-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F in each 0.5 mL dose.
  Arms: Prevnar 13™

SUMMARY:
The purpose of this study is to 1) evaluate the safety and tolerability of V114 and 2) to compare the immune responses of the 15 serotypes contained in V114 with V114 versus Prevnar 13™. The primary hypotheses are that 1) V114 is noninferior to Prevnar 13™ as measured by the serotype specific opsonophagocytic activity (OPA) geometric mean titers (GMTs) for 13 shared serotypes at 30 days postvaccination and that 2) V114 is superior to Prevnar 13™ as measured by serotype-specific OPA GMTs for 2 unique serotypes in V114 at 30 days postvaccination.

ELIGIBILITY:
Inclusion Criteria:

* Participant has good health in the opinion of the investigator. Any underlying chronic condition must be documented to be in stable condition according to the investigator's judgment.
* Male or female ≥50 years of age at the time of signing the informed consent. (For Japan only: Is male or female ≥65 years of age at the time of signing the informed consent)
* Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Female participant is eligible to participate if she is not pregnant, not breastfeeding, and is not a woman of childbearing potential (WOCBP) OR a WOCBP who agrees to use agreed upon contraception during the treatment period and for at least 6 weeks after the last dose of study intervention.
* Provides written informed consent for the study. The participant may also provide consent for future biomedical research. However, the participant may participate in the main study without participating in future biomedical research.

Exclusion Criteria:

* History of invasive pneumococcal disease (IPD) (positive blood culture, positive cerebrospinal fluid culture, or positive culture at another sterile site) or known history of other culture-positive pneumococcal disease within 3 years of Visit 1 (Day 1).
* Known hypersensitivity to any component of pneumococcal polysaccharide vaccine, pneumococcal conjugate vaccine (PCV), or any diphtheria toxoid-containing vaccine.
* Known or suspected impairment of immunological function including, but not limited to, a history of congenital or acquired immunodeficiency, documented human immunodeficiency virus (HIV) infection, functional or anatomic asplenia, or history of autoimmune disease.
* Coagulation disorder contraindicating intramuscular (IM) vaccinations.
* Recent febrile illness (defined as oral or tympanic temperature ≥100.4°F [≥38.0°C] or axillary or temporal temperature ≥99.4°F [≥37.4°C]) or received antibiotic therapy for any acute illness occurring within 72 hours before receipt of study vaccine.
* History of malignancy ≤5 years prior to signing informed consent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* A WOCBP who has a positive urine or serum pregnancy test before the first vaccination at Visit 1 (Day 1).
* Has received any pneumococcal vaccine or is expected to receive any pneumococcal vaccine during the study outside of the protocol.
* Has received systemic corticosteroids (prednisone equivalent of ≥20 mg/day) for ≥14 consecutive days and has not completed intervention at least 30 days before study entry.
* Has received systemic corticosteroids exceeding physiologic replacement doses (approximately 5 mg/day prednisone equivalent) within 14 days before vaccination. (Note: Topical, ophthalmic, intra-articular or soft-tissue [e.g., bursa, tendon steroid injections], and inhaled/nebulized steroids are permitted.)
* Is receiving immunosuppressive therapy, including chemotherapeutic agents used to treat cancer or other conditions, and interventions associated with organ or bone marrow transplantation, or autoimmune disease.
* Has received any non-live vaccine within the 14 days before receipt of any study vaccine or is scheduled to receive any non-live vaccine within 30 days following receipt of any study vaccine. (Exception: Inactivated influenza vaccine may be administered but must be given at least 7 days before receipt of any study vaccine or at least 15 days after receipt of any study vaccine.)
* Has received any live vaccine within 30 days before receipt of any study vaccine or is scheduled to receive any live vaccine within 30 days following receipt of any study vaccine.
* Has received a blood transfusion or blood products, including immunoglobulin, within the 6 months before receipt of study vaccine or is scheduled to receive a blood transfusion or blood product within 30 days of receipt of study vaccine. Autologous blood transfusions are not considered an exclusion criterion.
* Currently participating in or has participated in an interventional clinical study with an investigational compound or device within 2 months of participating in this current study.
* In the opinion of the investigator, has a history of clinically relevant drug or alcohol use that would interfere with participation in protocol-specified activities.
* History or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might expose the participant to risk by participating in the study, confound the results of the study, or interfere with the participant's participation for the full duration of the study.
* An immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is investigational site or Sponsor staff directly involved with this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1205 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (30):
- United States (14):
  - Synexus ( Site 1001), Mesa, Arizona
  - Artemis Institute for Clinical Research ( Site 1012), San Diego, California
  - Indago Research & Health Center, Inc ( Site 1002), Hialeah, Florida
  - Research Centers of America, LLC ( Site 1014), Hollywood, Florida
  - Advanced Medical Research Institute ( Site 0117), Miami, Florida
  - Lakes Research LLC ( Site 1005), Miami Lakes, Florida
  - Alliance for Multispecialty Research, LLC ( Site 1008), Newton, Kansas
  - Wake Research Clinical Research Center of Nevada, LLC ( Site 1010), Las Vegas, Nevada
  - Rapid Medical Research, Inc. ( Site 1011), Cleveland, Ohio
  - Diagnostics Research Group ( Site 1000), San Antonio, Texas
  - Synexus ( Site 1009), San Antonio, Texas
  - J Lewis Research Inc / Foothill Family Clinic ( Site 1013), Salt Lake City, Utah
  - Charlottesville Medical Research Center, LLC ( Site 1003), Charlottesville, Virginia
  - Health Research of Hampton Roads, Inc. ( Site 1007), Newport News, Virginia
- Canada (6):
  - Colchester Research Group ( Site 2002), Truro, Nova Scotia
  - Milestone Research ( Site 2003), London, Ontario
  - Bluewater Clinical Research Group Inc ( Site 2004), Sarnia, Ontario
  - Manna Research Inc.. ( Site 2007), Toronto, Ontario
  - Dynamik Research ( Site 2000), Pointe-Claire, Quebec
  - Q & T Research Sherbrooke Inc. ( Site 2001), Sherbrooke, Quebec
- Japan (5):
  - P-One Clinic, Keikokai Medical Corp. ( Site 0400), Hachiōji, Tokyo
  - Souseikai PS Clinic ( Site 0402), Fukuoka
  - Souseikai Nishikumamoto Hospital ( Site 0404), Kumamoto
  - Medical Corporation Heishinkai OPHAC Hospital ( Site 0401), Osaka
  - Medical Corporation Houeikai Sekino Clinical Pharmacology Clinic ( Site 0403), Tokyo
- Spain (3):
  - Hospital Universitario Quiron Madrid ( Site 0304), Pozuelo de Alarcón, Madrid
  - Instituto de Ciencias Medicas - ICM ( Site 0300), Alicante
  - CAP Centelles ( Site 0301), Centelles
- Taiwan (2):
  - National Cheng Kung University Hospital ( Site 0501), Dawan
  - National Taiwan University Hospital ( Site 0500), Taipei

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Platt HL, Cardona JF, Haranaka M, Schwartz HI, Narejos Perez S, Dowell A, Chang CJ, Dagan R, Tamms GM, Sterling T, Morgan L, Shi Y, Pedley A, Musey LK, Buchwald UK. A phase 3 trial of safety, tolerability, and immunogenicity of V114, 15-valent pneumococcal conjugate vaccine, compared with 13-valent pneumococcal conjugate vaccine in adults 50 years of age and older (PNEU-AGE). Vaccine. 2022 Jan 3;40(1):162-172. doi: 10.1016/j.vaccine.2021.08.049. Epub 2021 Sep 8. PMID 34507861

RESULTS

PARTICIPANT FLOW:
Groups:
- V114: Participants received a single 0.5 mL intramuscular (IM) injection of V114 on Day 1.
- Prevnar 13™: Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1.
Period: Overall Study
Arm/Group | V114 | Prevnar 13™
Started | 604 | 601
Vaccinated | 602 | 600
Completed | 596 | 594
Not Completed | 8 | 7
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Deviation | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 5 | 5
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V114 | Prevnar 13™ | Total
Number analyzed (Participants) | 604 | 601 | 1205
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.2 (7.7) | 65.7 (7.4) | 65.9 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 359 | 332 | 691
  Male | 245 | 269 | 514
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 135 | 129 | 264
  Not Hispanic or Latino | 469 | 471 | 940
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 150 | 152 | 302
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 36 | 37 | 73
  White | 410 | 407 | 817
  More than one race | 7 | 4 | 11
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Solicited Injection-site Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited injection-site AEs consist of redness/erythema, swelling, and tenderness/pain.
Time Frame: Up to Day 5 postvaccination
Population: The analysis population included all randomized participants who received study vaccination and were included in the intervention group according to the intervention they received.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 602 | 600
Percentage of Participants
  Injection site erythema | 9.0 | 11.3
  Injection site pain | 54.0 | 42.3
  Injection site swelling | 12.5 | 11.2
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Injection site redness/erythema; Test type: Other — Estimated differences, confidence intervals (CIs), and p-values are calculated based on the Miettinen & Nurminen method and are provided in accordance with the statistical analysis plan; p = 0.175, Miettinen & Nurminen; Difference in Percent = -2.4, 95% CI 2-sided [-5.8 to 1.1]
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Injection site tenderness/pain; Test type: Other — Estimated differences, CIs, and p-values are calculated based on the Miettinen & Nurminen method and are provided in accordance with the statistical analysis plan; p < 0.001, Miettinen & Nurminen; Difference in Percent = 11.7, 95% CI 2-sided [6.0 to 17.2]
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Injection site swelling; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.488, Miettinen & Nurminen; Difference in Percent = 1.3, 95% CI 2-sided [-2.4 to 5.0]

2. Primary Outcome: Percentage of Participants With Solicited Systemic Adverse Events
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following vaccination with V114 or Prevnar 13™, the percentage of participants with solicited systemic AEs was assessed. The solicited systemic AEs assessed were muscle pain/myalgia, joint pain/arthralgia, headache, and tiredness/fatigue.
Time Frame: Up to Day 14 postvaccination
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 602 | 600
Percentage of Participants
  Joint pain/arthralgia | 5.3 | 5.5
  Tiredness/fatigue | 17.4 | 17.3
  Headache | 11.6 | 13.0
  Muscle pain/myalgia | 15.4 | 12.0
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Joint pain/arthralgia; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.888, Miettinen & Nurminen; Difference in Percent = -0.2, 95% CI 2-sided [-2.8 to 2.4]
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Tiredness/fatigue; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.960, Miettinen & Nurminen; Difference in Percent = 0.1, 95% CI 2-sided [-4.2 to 4.4]
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Headache; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.469, Miettinen & Nurminen; Difference in Percent = -1.4, 95% CI 2-sided [-5.1 to 2.4]
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; Muscle pain/myalgia; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.082, Miettinen & Nurminen; Difference in Percent = 3.4, 95% CI 2-sided [-0.4 to 7.4]

3. Primary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event
Description: A serious adverse event (SAE) is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires inpatient hospitalization or prolongs existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is another important medical event. SAEs that are reported to be at least possibly related by the investigator to study vaccination will be summarized.
Time Frame: Up to Month 6
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 602 | 600
Percentage of Participants | 0.0 | 0.0
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Vaccine-related SAEs; Test type: Other — Estimated differences and CIs are calculated based on the Miettinen & Nurminen method and are provided in accordance with the statistical analysis plan; Miettinen & Nurminen; Difference in Percent = 0.0, 95% CI 2-sided [-0.6 to 0.6]

4. Primary Outcome: Geometric Mean Titer of Serotype-specific Opsonophagocytic Activity at Day 30
Description: Serotype-specific opsonophagocytic activity (OPA) geometric mean titers (GMTs) (estimated) and GMT ratios with 95% CIs and 1-sided p-values were calculated using a constrained longitudinal data analysis (cLDA) model utilizing data from both vaccination groups. Per the statistical analysis plan, the only CIs calculated were the between-group CIs (for the GMT ratios); within-group CIs were not calculated. OPA for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) were determined using a multiplexed opsonophagocytic assay (MOPA). The measure type of "number" presented in the data table below for serotype-specific OPA titer is the geometric mean.
Time Frame: Day 30
Population: The analysis population included all randomized participants without protocol deviations, such as failure to receive study vaccine or receipt of prohibited medication prior to study vaccination.
Measure: Number; unit: Titers
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 602 | 600
Titers
  Serotype 1 (Shared): number analyzed (Participants) | 598 | 598
  Serotype 1 (Shared) | 256.3 | 322.6
  Serotype 3 (Shared): number analyzed (Participants) | 598 | 598
  Serotype 3 (Shared) | 216.2 | 135.1
  Serotype 4 (Shared): number analyzed (Participants) | 598 | 598
  Serotype 4 (Shared) | 1125.6 | 1661.6
  Serotype 5 (Shared): number analyzed (Participants) | 598 | 598
  Serotype 5 (Shared) | 447.3 | 563.5
  Serotype 6A (Shared): number analyzed (Participants) | 596 | 598
  Serotype 6A (Shared) | 5407.2 | 5424.5
  Serotype 6B (Shared): number analyzed (Participants) | 598 | 598
  Serotype 6B (Shared) | 4011.7 | 3258.2
  Serotype 7F (Shared): number analyzed (Participants) | 597 | 598
  Serotype 7F (Shared) | 4617.3 | 5880.6
  Serotype 9V (Shared): number analyzed (Participants) | 598 | 597
  Serotype 9V (Shared) | 1817.3 | 2232.9
  Serotype 14 (Shared): number analyzed (Participants) | 598 | 598
  Serotype 14 (Shared) | 1999.3 | 2656.7
  Serotype 18C (Shared): number analyzed (Participants) | 598 | 598
  Serotype 18C (Shared) | 2757.7 | 2583.7
  Serotype 19A (Shared): number analyzed (Participants) | 598 | 598
  Serotype 19A (Shared) | 3194.3 | 3979.8
  Serotype 19F (Shared): number analyzed (Participants) | 598 | 598
  Serotype 19F (Shared) | 1695.1 | 1917.8
  Serotype 23F (Shared): number analyzed (Participants) | 598 | 598
  Serotype 23F (Shared) | 2045.4 | 1740.4
  Serotype 22F (Unique to V114): number analyzed (Participants) | 594 | 586
  Serotype 22F (Unique to V114) | 2375.2 | 74.6
  Serotype 33F (Unique to V114): number analyzed (Participants) | 598 | 597
  Serotype 33F (Unique to V114) | 7994.7 | 1124.9
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Serotype 1 (Shared); Test type: Non-Inferiority — The statistical criterion for noninferiority requires the lower bound of the 2-sided 95% confidence interval (CI) of the OPA GMT ratio (V114/ Prevnar 13™) to be greater than 0.5; p < 0.001, Constrained longitudinal data analysis; GMT ratio, 95% CI, and p-value are estimated from a constrained longitudinal data analysis (cLDA) model; GMT Ratio = 0.79, 95% CI 2-sided [0.66 to 0.96]
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Serotype 3 (Shared); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI, and p-value are estimated from a cLDA model; GMT Ratio = 1.60, 95% CI 2-sided [1.38 to 1.85]
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Serotype 4 (Shared); Test type: Non-Inferiority — The statistical criterion for noninferiority requires the lower bound of the 2-sided 95% CI of the OPA GMT ratio (V114/ Prevnar 13™) to be greater than 0.5; p < 0.001, cLDA; GMT ratio, 95% CI, and p-value are estimated from a cLDA model; GMT Ratio = 0.68, 95% CI 2-sided [0.57 to 0.80]
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; Serotype 5 (Shared); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI, and p-value are estimated from a cLDA model; GMT Ratio = 0.79, 95% CI 2-sided [0.64 to 0.98]
Statistical Analysis 5: Comparison: V114 vs Prevnar 13™; Serotype 6A (Shared); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI, and p-value are estimated from a cLDA model; GMT Ratio = 1.00, 95% CI 2-sided [0.84 to 1.19]
Statistical Analysis 6: Comparison: V114 vs Prevnar 13™; Serotype 6B (Shared); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI, and p-value are estimated from a cLDA model; GMT Ratio = 1.23, 95% CI 2-sided [1.02 to 1.48]
Statistical Analysis 7: Comparison: V114 vs Prevnar 13™; Serotype 7F (Shared); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI, and p-value are estimated from a cLDA model; GMT Ratio = 0.79, 95% CI 2-sided [0.68 to 0.90]
Statistical Analysis 8: Comparison: V114 vs Prevnar 13™; Serotype 9V (Shared); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI, and p-value are estimated from a cLDA model; GMT Ratio = 0.81, 95% CI 2-sided [0.70 to 0.94]
Statistical Analysis 9: Comparison: V114 vs Prevnar 13™; Serotype 14 (Shared); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI, and p-value are estimated from a cLDA model; GMT Ratio = 0.75, 95% CI 2-sided [0.64 to 0.89]
Statistical Analysis 10: Comparison: V114 vs Prevnar 13™; Serotype 18C (Shared); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI, and p-value are estimated from a cLDA model; GMT Ratio = 1.07, 95% CI 2-sided [0.91 to 1.26]
Statistical Analysis 11: Comparison: V114 vs Prevnar 13™; Serotype 19A (Shared); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI, and p-value are estimated from a cLDA model; GMT Ratio = 0.80, 95% CI 2-sided [0.70 to 0.93]
Statistical Analysis 12: Comparison: V114 vs Prevnar 13™; Serotype 19F (Shared); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI, and p-value are estimated from a cLDA model; GMT Ratio = 0.88, 95% CI 2-sided [0.76 to 1.02]
Statistical Analysis 13: Comparison: V114 vs Prevnar 13™; Serotype 23F (Shared); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, cLDA; GMT ratio, 95% CI, and p-value are estimated from a cLDA model; GMT Ratio = 1.18, 95% CI 2-sided [0.96 to 1.44]
Statistical Analysis 14: Comparison: V114 vs Prevnar 13™; Serotype 22F (Unique to V114); Test type: Superiority — The statistical criterion for superiority requires the lower bound of the 2-sided 95% CI of the OPA GMT ratio [V114/ Prevnar 13™] to be greater than 2.0; p < 0.001, cLDA; GMT ratio, 95% CI, and p-value are estimated from a cLDA model; GMT Ratio = 31.83, 95% CI 2-sided [25.35 to 39.97]
Statistical Analysis 15: Comparison: V114 vs Prevnar 13™; Serotype 33F (Unique to V114); Test type: Superiority — [test comment as in outcome 4, analysis 14]; p < 0.001, cLDA; GMT ratio, 95% CI, and p-value are estimated from a cLDA model; GMT Ratio = 7.11, 95% CI 2-sided [6.07 to 8.32]

5. Primary Outcome: Percentage of Participants With ≥4 Fold Rise in Serotype-specific OPA for 2 Unique V114 Serotypes
Description: Activity for the serotypes contained in Prevnar 13™ and V114 was determined using a multiplexed opsonophagocytic assay (MOPA). The percentage of participants who had ≥4-fold rise in OPA titers were calculated from baseline (Day 1) to 30 days postvaccination (Day 30) for OPA responses for the 2 unique serotypes in V114. The observed response percentage (m/n) included: m=the number of participants with the indicated response divided by n=the number of participants contributing to the analysis. Per the statistical analysis plan, the only CIs calculated were the between-group CIs (for the percentage point difference); within-group CIs were not calculated.
Time Frame: Day 1 (Baseline) and Day 30
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 602 | 600
Percentage of Participants
  Serotype 22F (Unique to V114): number analyzed (Participants) | 524 | 498
  Serotype 22F (Unique to V114) | 71.4 | 14.3
  Serotype 33F (Unique to V114): number analyzed (Participants) | 578 | 560
  Serotype 33F (Unique to V114) | 56.7 | 6.3
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Serotype 22F (Unique to V114); Test type: Superiority — The statistical criterion for superiority requires the lower bound of the 2-sided 95% CI of the differences [V114 - Prevnar 13™] between the proportions of participants with a ≥4-fold rise from prevaccination [Day 1] to 30 days postvaccination [Day 30] to be greater than 0.1; p < 0.001, Miettinen & Nurminen; Estimated difference, 95% CI, and p-value are based on the stratified Miettinen & Nurminen method; Percentage Point Difference = 57.1, 95% CI 2-sided [52.0 to 61.8]
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Serotype 33F (Unique to V114); Test type: Superiority — The statistical criterion for superiority requires the lower bound of the 2-sided 95% CI of the differences [V114 - Prevnar 13™] between the proportions of participants with a ≥4-fold rise from prevaccination [Day 1] to 30 days postvaccination [Day 30] to be greater than 0.1); p < 0.001, Miettinen & Nurminen; Estimated difference, 95% CI, and p-value are based on the stratified Miettinen & Nurminen method; Percentage Point Difference = 50.5, 95% CI 2-sided [45.9 to 54.9]

6. Secondary Outcome: GMT of Serotype-specific OPA for Serotype 3 at Day 30
Description: Serotype-specific OPA GMTs (estimated) and GMT ratios with 95% CIs and 1-sided p-values were calculated using a cLDA model utilizing data from both vaccination groups. Per the statistical analysis plan, the only CIs calculated were the between-group CIs (for the GMT ratios); within-group CIs were not calculated. OPA for serotype 3 contained in Prevnar 13™ and V114 was determined using a MOPA. The measure type of "number" presented in the data table below for serotype-specific OPA titer is the geometric mean.
Time Frame: Day 30
Population: as for outcome 4
Measure: Number; unit: Titers
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 598 | 598
Titers | 216.2 | 135.1
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Serotype 3 (Shared); Test type: Superiority — The statistical criterion for superiority requires the lower bound of the 2-sided 95% CI of the OPA GMT ratio [V114/ Prevnar 13™] to be greater than 1.2; p < 0.001, cLDA; GMT ratio, 95% CI, and p-value are estimated from a cLDA model; GMT Ratio = 1.60, 95% CI 2-sided [1.38 to 1.85]

7. Secondary Outcome: Percentage of Participants With ≥4 Fold Rise in Serotype-specific OPA for Serotype 3 OPA Responses
Description: Activity for serotype 3 contained in Prevnar 13™ and V114 was determined using a MOPA. The observed response percentage of participants (m/n) who had ≥4-fold rise in OPA titers were calculated from baseline to postvaccination. n=Number of participants contributing to the analysis; m=Number of participants with the indicated response. Per the statistical analysis plan, the only CIs calculated were the between-group CIs (for the percentage point difference); within-group CIs were not calculated.
Time Frame: Day 1 (Baseline) and Day 30
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 580 | 576
Percentage of Participants | 70.2 | 58.7
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Serotype 3 (Shared) ≥4-Fold Rise in OPA; Test type: Superiority — The statistical criterion for superiority requires the lower bound of the 2-sided 95% CI of the difference(V114 - Prevnar 13™) between the proportions of participants with a ≥4-fold rise from prevaccination (Day 1) to 30 days postvaccination (Day 30) to be greater than 0; p < 0.001, Miettinen & Nurminen; Estimated difference, 95% CI, and p-value are based on the stratified Miettinen & Nurminen method; Percentage Point Difference = 11.5, 95% CI 2-sided [6.0 to 16.9]

8. Secondary Outcome: Geometric Mean Concentration of Serotype-specific IgG at Day 30
Description: Serotype-specific Immunoglobulin G (IgG) geometric mean concentrations (GMCs) (estimated) and GMC ratios with 95% confidence intervals (CIs) and 1-sided p-values were calculated using a cLDA model utilizing data from both vaccination groups. Per the statistical analysis plan, the only CIs calculated were the between-group CIs (for the GMC ratios); within-group CIs were not calculated. IgG for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) will be determined using an electrochemiluminescence assay. The measure type of "number" presented in the data table below for serotype-specific IgG concentration is the geometric mean.
Time Frame: Day 30
Population: as for outcome 4
Measure: Number; unit: µg/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 602 | 600
µg/mL
  Serotype 1 (Shared): number analyzed (Participants) | 598 | 598
  Serotype 1 (Shared) | 5.30 | 7.34
  Serotype 3 (Shared): number analyzed (Participants) | 598 | 598
  Serotype 3 (Shared) | 0.96 | 0.64
  Serotype 4 (Shared): number analyzed (Participants) | 598 | 598
  Serotype 4 (Shared) | 1.88 | 2.62
  Serotype 5 (Shared): number analyzed (Participants) | 598 | 598
  Serotype 5 (Shared) | 4.57 | 5.56
  Serotype 6A (Shared): number analyzed (Participants) | 598 | 598
  Serotype 6A (Shared) | 7.21 | 7.01
  Serotype 6B (Shared): number analyzed (Participants) | 598 | 598
  Serotype 6B (Shared) | 8.60 | 6.19
  Serotype 7F (Shared): number analyzed (Participants) | 598 | 598
  Serotype 7F (Shared) | 6.18 | 8.09
  Serotype 9V (Shared): number analyzed (Participants) | 598 | 598
  Serotype 9V (Shared) | 4.77 | 5.52
  Serotype 14 (Shared): number analyzed (Participants) | 598 | 598
  Serotype 14 (Shared) | 9.39 | 12.30
  Serotype 18C (Shared): number analyzed (Participants) | 598 | 598
  Serotype 18C (Shared) | 8.99 | 10.00
  Serotype 19A (Shared): number analyzed (Participants) | 598 | 598
  Serotype 19A (Shared) | 14.60 | 17.38
  Serotype 19F (Shared): number analyzed (Participants) | 598 | 598
  Serotype 19F (Shared) | 8.77 | 9.70
  Serotype 23F (Shared): number analyzed (Participants) | 598 | 598
  Serotype 23F (Shared) | 6.67 | 6.13
  Serotype 22F (Unique to V114): number analyzed (Participants) | 598 | 598
  Serotype 22F (Unique to V114) | 3.44 | 0.32
  Serotype 33F (Unique to V114): number analyzed (Participants) | 598 | 598
  Serotype 33F (Unique to V114) | 11.05 | 1.23
Statistical Analysis 1: Comparison: V114 vs Prevnar 13™; Serotype 1 (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a constrained longitudinal data analysis (cLDA) model; GMC Ratio = 0.72, 95% CI 2-sided [0.62 to 0.83]
Statistical Analysis 2: Comparison: V114 vs Prevnar 13™; Serotype 3 (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.51, 95% CI 2-sided [1.33 to 1.71]
Statistical Analysis 3: Comparison: V114 vs Prevnar 13™; Serotype 4 (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 0.72, 95% CI 2-sided [0.62 to 0.83]
Statistical Analysis 4: Comparison: V114 vs Prevnar 13™; Serotype 5 (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 0.82, 95% CI 2-sided [0.70 to 0.96]
Statistical Analysis 5: Comparison: V114 vs Prevnar 13™; Serotype 6A (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.03, 95% CI 2-sided [0.87 to 1.21]
Statistical Analysis 6: Comparison: V114 vs Prevnar 13™; Serotype 6B (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.39, 95% CI 2-sided [1.17 to 1.64]
Statistical Analysis 7: Comparison: V114 vs Prevnar 13™; Serotype 7F (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 0.76, 95% CI 2-sided [0.66 to 0.89]
Statistical Analysis 8: Comparison: V114 vs Prevnar 13™; Serotype 9V (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 0.86, 95% CI 2-sided [0.75 to 1.00]
Statistical Analysis 9: Comparison: V114 vs Prevnar 13™; Serotype 14 (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 0.76, 95% CI 2-sided [0.65 to 0.89]
Statistical Analysis 10: Comparison: V114 vs Prevnar 13™; Serotype 18C (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 0.90, 95% CI 2-sided [0.77 to 1.05]
Statistical Analysis 11: Comparison: V114 vs Prevnar 13™; Serotype 19A (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 0.84, 95% CI 2-sided [0.73 to 0.97]
Statistical Analysis 12: Comparison: V114 vs Prevnar 13™; Serotype 19F (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 0.90, 95% CI 2-sided [0.78 to 1.05]
Statistical Analysis 13: Comparison: V114 vs Prevnar 13™; Serotype 23F (Shared); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 1.09, 95% CI 2-sided [0.92 to 1.28]
Statistical Analysis 14: Comparison: V114 vs Prevnar 13™; Serotype 22F (Unique to V114); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 10.62, 95% CI 2-sided [9.37 to 12.03]
Statistical Analysis 15: Comparison: V114 vs Prevnar 13™; Serotype 33F (Unique to V114); Test type: Other — GMC ratio and 95% CI are estimated from a cLDA model; GMC Ratio = 8.98, 95% CI 2-sided [8.00 to 10.07]

9. Secondary Outcome: Geometric Mean Fold Rise in Serotype-specific OPA
Description: Activity for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using a Multiplexed Opsonophagocytic Assay. Geometric mean fold rise (GMFR) is defined as the geometric mean of the ratio of concentration at Day 30 after vaccination divided by concentration at baseline.
Time Frame: Day 1 (Baseline) and Day 30
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 602 | 600
Ratio
  Serotype 1 (Shared): number analyzed (Participants) | 583 | 573
  Serotype 1 (Shared) | 14.3 [12.5 to 16.4] | 18.7 [16.2 to 21.5]
  Serotype 3 (Shared): number analyzed (Participants) | 580 | 576
  Serotype 3 (Shared) | 7.7 [7.0 to 8.6] | 5.2 [4.7 to 5.7]
  Serotype 4 (Shared): number analyzed (Participants) | 586 | 578
  Serotype 4 (Shared) | 17.8 [15.7 to 20.3] | 24.4 [21.3 to 27.8]
  Serotype 5 (Shared): number analyzed (Participants) | 588 | 584
  Serotype 5 (Shared) | 12.3 [10.7 to 14.2] | 15.3 [13.2 to 17.6]
  Serotype 6A (Shared): number analyzed (Participants) | 545 | 550
  Serotype 6A (Shared) | 13.0 [11.4 to 14.9] | 13.3 [11.6 to 15.2]
  Serotype 6B (Shared): number analyzed (Participants) | 579 | 576
  Serotype 6B (Shared) | 26.3 [22.4 to 30.8] | 21.6 [18.5 to 25.2]
  Serotype 7F (Shared): number analyzed (Participants) | 566 | 555
  Serotype 7F (Shared) | 12.0 [10.3 to 13.9] | 14.1 [12.1 to 16.5]
  Serotype 9V (Shared): number analyzed (Participants) | 578 | 573
  Serotype 9V (Shared) | 5.3 [4.8 to 6.0] | 6.3 [5.6 to 7.1]
  Serotype 14 (Shared): number analyzed (Participants) | 579 | 576
  Serotype 14 (Shared) | 6.2 [5.4 to 7.2] | 8.7 [7.5 to 10.0]
  Serotype 18C (Shared): number analyzed (Participants) | 578 | 579
  Serotype 18C (Shared) | 11.3 [10.0 to 12.9] | 10.4 [9.1 to 11.8]
  Serotype 19A (Shared): number analyzed (Participants) | 581 | 575
  Serotype 19A (Shared) | 10.9 [9.5 to 12.5] | 13.1 [11.4 to 15.1]
  Serotype 19F (Shared): number analyzed (Participants) | 579 | 576
  Serotype 19F (Shared) | 6.6 [5.9 to 7.5] | 7.4 [6.6 to 8.3]
  Serotype 23F (Shared): number analyzed (Participants) | 555 | 555
  Serotype 23F (Shared) | 16.2 [14.0 to 18.9] | 13.5 [11.5 to 15.9]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 524 | 498
  Serotype 22F (Unique to V114) | 28.3 [22.8 to 35.1] | 1.2 [1.0 to 1.4]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 578 | 560
  Serotype 33F (Unique to V114) | 7.4 [6.4 to 8.6] | 1.0 [1.0 to 1.2]

10. Secondary Outcome: Geometric Mean Fold Rise in Serotype-specific IgG
Description: Activity for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using an electrochemiluminescence assay. Geometric mean fold rise (GMFR) is defined as the geometric mean of the ratio of concentration at Day 30 after vaccination divided by concentration at baseline.
Time Frame: Day 1 (Baseline) and Day 30
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 602 | 600
Ratio
  Serotype 1 (Shared): number analyzed (Participants) | 588 | 584
  Serotype 1 (Shared) | 10.6 [9.4 to 12.0] | 14.7 [13.1 to 16.6]
  Serotype 3 (Shared): number analyzed (Participants) | 588 | 582
  Serotype 3 (Shared) | 6.8 [6.2 to 7.6] | 4.7 [4.2 to 5.1]
  Serotype 4 (Shared): number analyzed (Participants) | 586 | 583
  Serotype 4 (Shared) | 8.0 [7.2 to 9.0] | 11.2 [10.0 to 12.5]
  Serotype 5 (Shared): number analyzed (Participants) | 588 | 584
  Serotype 5 (Shared) | 4.7 [4.2 to 5.2] | 5.8 [5.2 to 6.5]
  Serotype 6A (Shared): number analyzed (Participants) | 588 | 584
  Serotype 6A (Shared) | 19.9 [17.6 to 22.6] | 19.7 [17.4 to 22.3]
  Serotype 6B (Shared): number analyzed (Participants) | 588 | 582
  Serotype 6B (Shared) | 19.1 [16.8 to 21.7] | 13.8 [12.3 to 15.6]
  Serotype 7F (Shared): number analyzed (Participants) | 588 | 584
  Serotype 7F (Shared) | 12.3 [10.9 to 13.9] | 15.8 [13.9 to 18.0]
  Serotype 9V (Shared): number analyzed (Participants) | 588 | 584
  Serotype 9V (Shared) | 9.9 [8.9 to 11.1] | 11.1 [9.9 to 12.4]
  Serotype 14 (Shared): number analyzed (Participants) | 587 | 583
  Serotype 14 (Shared) | 5.1 [4.5 to 5.7] | 7.2 [6.3 to 8.2]
  Serotype 18C (Shared): number analyzed (Participants) | 588 | 583
  Serotype 18C (Shared) | 12.8 [11.3 to 14.5] | 14.3 [12.6 to 16.2]
  Serotype 19A (Shared): number analyzed (Participants) | 588 | 584
  Serotype 19A (Shared) | 8.7 [7.8 to 9.8] | 10.6 [9.5 to 11.9]
  Serotype 19F (Shared): number analyzed (Participants) | 583 | 580
  Serotype 19F (Shared) | 10.9 [9.7 to 12.3] | 12.5 [11.1 to 14.0]
  Serotype 23F (Shared): number analyzed (Participants) | 586 | 584
  Serotype 23F (Shared) | 13.5 [11.9 to 15.3] | 12.2 [10.8 to 13.7]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 588 | 583
  Serotype 22F (Unique to V114) | 11.7 [10.3 to 13.3] | 1.1 [1.1 to 1.1]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 588 | 584
  Serotype 33F (Unique to V114) | 9.1 [8.0 to 10.2] | 1.0 [1.0 to 1.0]

11. Secondary Outcome: Percentage of Participants With ≥4-Fold Rise in Serotype-specific OPA Titer
Description: Activity for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) was determined using a multiplexed opsonophagocytic assay. The percentage of participants who had ≥4-fold rise in OPA titers were calculated from baseline to postvaccination.
Time Frame: Day 1 (Baseline) and Day 30
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 602 | 600
Percentage of Participants
  Serotype 1 (Shared): number analyzed (Participants) | 583 | 573
  Serotype 1 (Shared) | 75.1 [71.4 to 78.6] | 77.7 [74.0 to 81.0]
  Serotype 3 (Shared): number analyzed (Participants) | 580 | 576
  Serotype 3 (Shared) | 70.2 [66.3 to 73.9] | 58.7 [54.5 to 62.7]
  Serotype 4 (Shared): number analyzed (Participants) | 586 | 578
  Serotype 4 (Shared) | 79.5 [76.0 to 82.7] | 84.8 [81.6 to 87.6]
  Serotype 5 (Shared): number analyzed (Participants) | 588 | 584
  Serotype 5 (Shared) | 71.6 [67.8 to 75.2] | 75.3 [71.6 to 78.8]
  Serotype 6A (Shared): number analyzed (Participants) | 545 | 550
  Serotype 6A (Shared) | 76.5 [72.7 to 80.0] | 74.9 [71.1 to 78.5]
  Serotype 6B (Shared): number analyzed (Participants) | 579 | 576
  Serotype 6B (Shared) | 81.2 [77.7 to 84.3] | 79.2 [75.6 to 82.4]
  Serotype 7F (Shared): number analyzed (Participants) | 566 | 555
  Serotype 7F (Shared) | 66.4 [62.4 to 70.3] | 72.4 [68.5 to 76.1]
  Serotype 9V (Shared): number analyzed (Participants) | 578 | 573
  Serotype 9V (Shared) | 54.0 [49.8 to 58.1] | 60.0 [55.9 to 64.1]
  Serotype 14 (Shared): number analyzed (Participants) | 579 | 576
  Serotype 14 (Shared) | 52.2 [48.0 to 56.3] | 60.8 [56.6 to 64.8]
  Serotype 18C (Shared): number analyzed (Participants) | 578 | 579
  Serotype 18C (Shared) | 71.3 [67.4 to 74.9] | 69.1 [65.1 to 72.8]
  Serotype 19A (Shared): number analyzed (Participants) | 581 | 575
  Serotype 19A (Shared) | 70.6 [66.7 to 74.2] | 71.1 [67.2 to 74.8]
  Serotype 19F (Shared): number analyzed (Participants) | 579 | 576
  Serotype 19F (Shared) | 62.0 [57.9 to 66.0] | 65.1 [61.1 to 69.0]
  Serotype 23F (Shared): number analyzed (Participants) | 555 | 555
  Serotype 23F (Shared) | 75.0 [71.1 to 78.5] | 71.4 [67.4 to 75.1]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 524 | 498
  Serotype 22F (Unique to V114) | 71.4 [67.3 to 75.2] | 14.3 [11.3 to 17.6]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 578 | 560
  Serotype 33F (Unique to V114) | 56.7 [52.6 to 60.8] | 6.3 [4.4 to 8.6]

12. Secondary Outcome: Percentage of Participants With ≥4-Fold Rise in Serotype-specific IgG Concentration
Description: Activity for the serotypes contained in Prevnar 13™ and V114 (13 serotypes shared with Prevnar 13™ and 2 serotypes unique to V114) will be determined using an electrochemiluminescence assay. The percentage of participants who had ≥4-fold rise in IgG concentration are calculated from baseline to postvaccination.
Time Frame: Day 1 (Baseline) and Day 30
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 602 | 600
Percentage of Participants
  Serotype 1 (Shared): number analyzed (Participants) | 588 | 584
  Serotype 1 (Shared) | 73.1 [69.4 to 76.7] | 78.4 [74.9 to 81.7]
  Serotype 3 (Shared): number analyzed (Participants) | 588 | 582
  Serotype 3 (Shared) | 61.6 [57.5 to 65.5] | 51.4 [47.2 to 55.5]
  Serotype 4 (Shared): number analyzed (Participants) | 586 | 583
  Serotype 4 (Shared) | 65.0 [61.0 to 68.9] | 76.0 [72.3 to 79.4]
  Serotype 5 (Shared): number analyzed (Participants) | 588 | 584
  Serotype 5 (Shared) | 45.1 [41.0 to 49.2] | 53.4 [49.3 to 57.5]
  Serotype 6A (Shared): number analyzed (Participants) | 588 | 584
  Serotype 6A (Shared) | 83.5 [80.3 to 86.4] | 83.4 [80.1 to 86.3]
  Serotype 6B (Shared): number analyzed (Participants) | 588 | 582
  Serotype 6B (Shared) | 82.8 [79.5 to 85.8] | 77.5 [73.9 to 80.8]
  Serotype 7F (Shared): number analyzed (Participants) | 588 | 584
  Serotype 7F (Shared) | 73.5 [69.7 to 77.0] | 78.6 [75.0 to 81.9]
  Serotype 9V (Shared): number analyzed (Participants) | 588 | 584
  Serotype 9V (Shared) | 69.6 [65.7 to 73.3] | 75.5 [71.8 to 79.0]
  Serotype 14 (Shared): number analyzed (Participants) | 587 | 583
  Serotype 14 (Shared) | 49.4 [45.3 to 53.5] | 59.5 [55.4 to 63.5]
  Serotype 18C (Shared): number analyzed (Participants) | 588 | 583
  Serotype 18C (Shared) | 73.1 [69.4 to 76.7] | 76.3 [72.7 to 79.7]
  Serotype 19A (Shared): number analyzed (Participants) | 588 | 584
  Serotype 19A (Shared) | 67.2 [63.2 to 71.0] | 71.2 [67.4 to 74.9]
  Serotype 19F (Shared): number analyzed (Participants) | 583 | 580
  Serotype 19F (Shared) | 69.5 [65.6 to 73.2] | 75.5 [71.8 to 79.0]
  Serotype 23F (Shared): number analyzed (Participants) | 586 | 584
  Serotype 23F (Shared) | 74.9 [71.2 to 78.4] | 74.3 [70.6 to 77.8]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 588 | 583
  Serotype 22F (Unique to V114) | 71.4 [67.6 to 75.0] | 1.7 [0.8 to 3.1]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 588 | 584
  Serotype 33F (Unique to V114) | 66.5 [62.5 to 70.3] | 1.7 [0.8 to 3.1]

ADVERSE EVENTS:
Time Frame: Non-serious adverse events: Up to 14 days after vaccination; Serious adverse events and all-cause mortality: Up to ~Month 6 (Up to 194 days after vaccination).
Description: The analysis population for adverse events and serious adverse events: all randomized participants who received study vaccination and were included in the intervention group according to the intervention they received. The analysis population for the all cause mortality: all randomized participants.
Groups:
- PCV13: Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1.
Arm/Group | V114 | PCV13
All-Cause Mortality (participants affected / at risk) | 1/604 | 1/601
Serious Adverse Events (participants affected / at risk) | 9/602 | 13/600
Other Adverse Events (participants affected / at risk) | 395/602 | 336/600
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=602) | PCV13 (N=600)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=602) | PCV13 (N=600)
Fatigue (General disorders) | 105 (144) | 104 (140)
Injection site erythema (General disorders) | 60 (62) | 73 (77)
Injection site pain (General disorders) | 327 (367) | 257 (294)
Injection site swelling (General disorders) | 76 (79) | 73 (78)
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 (38) | 33 (39)
Myalgia (Musculoskeletal and connective tissue disorders) | 93 (111) | 72 (85)
Headache (Nervous system disorders) | 70 (93) | 78 (105)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT03950622/Prot_SAP_000.pdf